CLINICAL TRIAL: NCT01621100
Title: A Prospective, Open-Label, Multicenter, Single-Arm, Interventional Study to Evaluate the Efficacy and Tolerability of Once-Daily Oros Hydromorphone for Cancer Pain Treatment in Korean Cancer Patients.
Brief Title: Study to Evaluate Effectiveness and Tolerability of OROS Hydromorphone for Cancer Pain Treatment in Korean Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100659; HYD-KOR-4003 (Other: Janssen Korea, Ltd., Korea); 42801PAI4012 (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2012-04-10; First posted 2012-06-18 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: Cancer Pain
Keywords: Cancer pain; OROS; Osmotic release oral system; Hydromorphone; Painkiller; Opioid analgesic; Korean patients
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OROS hydromorphone (Experimental): Once-Daily OROS (Osmotic release oral system [a controlled release oral drug delivery system in the form of a tablet]) hydromorphone
  Interventions: Drug: OROS hydromorphone

INTERVENTIONS:
Drug: OROS hydromorphone — Type= exact number, unit= mg, number= 4, form= tablet, route= oral, administered from 1st evaluation day (Day 1) to 2nd evaluation day (Day 15±2). Dosage adjustment: If NRS (Numeric Rating Scale) =4 or more then dose can be increased by 4mg until the average pain intensity for the past 24 hours is adjusted to lower than NRS 3. For the treatment of breakthrough pain, if necessary the one-time administration dose of quick-effect OROS Hydromorphone shall be 2mg up to the daily dosage of the study medicine, 12mg.

SUMMARY:
The purpose of this study is to evaluate the effectiveness and tolerability of Once-Daily OROS ("Osmotic Release Oral System" [a controlled release oral medication delivery system in the form of a tablet]) hydromorphone for cancer pain treatment in Korean cancer patients.

DETAILED DESCRIPTION:
This is a prospective (expected to happen), open-label (type of clinical study in which both the researchers and participants know which treatment is being administered), multicenter (conducted at multiple centers), single-arm (only one group), study to evaluate the effectiveness and tolerability (capable to tolerate) of Once-Daily OROS hydromorphone for cancer pain treatment. This is a 14-week study consisting of 2-week efficacy evaluation period (1st evaluation on Day 1 and 2nd evaluation on Days 15±2) and a 12-week extension phase. 99 patients will receive Once-Daily OROS hydromorphone for 2 weeks .After 2 weeks, if a patient has continuous cancer pain and the investigator deems it necessary to administer the same medicine as the study medication then the patient may participate voluntarily in the 12 weeks extension phase. At the extension phase, other continuous-type strong opioid analgesics (painkiller) may be administered at the same time for the adjustment of cancer pain based on the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Cancer pain and require opioid analgesics
* Average pain intensity measured at the baseline (patient's medical status before any treatment or research is done) for the past 24 hours over Numeric Rating Scale (NRS) is 4
* Never taken continuous-type strong opioid analgesics
* Must be post-menopausal or if pre-menopausal, must use an acceptable method of birth control

Exclusion Criteria:

* Acute digestion related disease, such as dysphagia (difficulty in swallowing), vomiting, no enterokinesia (movements of intestine), intestinal obstruction, acute intestinal stricture (narrowing of a passageway)
* Expected to undergo radioactive treatment (radiation therapy) between Day 1 and Day 15 of study
* Being administered with monoamine oxidase inhibitor (eg, moclobemide, selegiline, toloxatone, etc) or within 2 weeks of administration thereof

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2011-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with 50% or more average Pain Intensity Difference (PID) from 1st evaluation day (Day 1) to the 2nd evaluation day (Days 15±2) | up to 17 days
  Average pain intensity is calculated (on 1st and 2nd evaluation days) for the past 24 hours of the patient using the NRS (Numeric Rating Scale) (0 = No pain, 10 = Unimaginably acute pain). PID (pain intensity difference) %= [NRS (1st evaluation day) - NRS (2nd evaluation day)]/ NRS (1st evaluation day).

SECONDARY OUTCOMES:
Korean Brief Pain Inventory (K-BPI) scores | up to 17 days
  A survey (questionnaire) to measures the pain intensity, the effect of pain on the performance of everyday life, effect of medicines for pain treatment and degree of pain reduction.
European Organization for Research and Treatment of Cancer Quality of Life (EORTC QLQ-C30) scores | up to 17 days
  Quality of life measurement survey with 30 questions that ask about the health status of cancer patients.
Patient's Global Assessment (PGA) scores | up to 17 days
  Patient checks any of the 5 stages: 1 = Not effective, 2 = Normal, 3 = Effective, 4 = Very Effective, 5 = Excellently effective based on how effective the study medication is in their treatment of pain after the last evaluation.
Investigator's Global Assessment scores | up to 17 days
  Study investigator checks any of the 5 stages: 1 = Not effective, 2 = Normal, 3 = Effective, 4 = Very Effective, 5 = Excellently effective based on how effective the study medication is in their treatment of pain after the last evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd Clinical Trial, Study Director — Janssen Korea, Ltd
Locations (6):
- South Korea (6):
  - Cheonan
  - Cheongju-si
  - Daejeon
  - Hwasun Gun
  - Jeonju
  - Jinju

REFERENCES:
- See also: A Prospective, Open-Label, Multicenter, Single-Arm, Interventional Study to Evaluate the Efficacy and Tolerability of Once-Daily Oros Hydromorphone for Cancer Pain Treatment in Korean Cancer Patients — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=3208&filename=CR100659_CSR.pdf